CLINICAL TRIAL: NCT01903603
Title: A Longitudinal Study of Movement and Participation in Patients With Cerebral Palsy: a Combined Brain Imaging and Kinematic Analysis
Brief Title: A Longitudinal Study of Movement and Participation in Patients With Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 100-4545A3; NSC101-2314-B-182-004-MY3 (Other: National Science Council)
Record Dates: First submitted 2013-07-17; First posted 2013-07-19 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2016-09

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; multi-modal brain techniques; MRI; Kinematic; motor control
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Healthy Children: Inclusion criteria for healthy children were as follows: ages of 4-20 y/o ; good cognition and cooperation; and healthy children.
- CP subjects: Inclusion criteria for subjects with brain damage by CP were as follows: a diagnosis of CP and aged 4-20 years old.

SUMMARY:
The primary goal of this study is to establish and evaluate an image-based biomarker for the impaired motor control and sensory information processing present in Cerebral palsy (CP) patients

DETAILED DESCRIPTION:
Cerebral palsy (CP) may lead to various motor deficits, which further influence the activities and participation. It would be ideal to characterize neural network and motor control model in patients with CP that underlies their clinical behavior by identifying altered neural network and motor control associated with behavioral improvement. The aim of this study is to investigate the brain image and motor control in patients with CP evaluated by multimodal imaging studies utilizing multi-modal techniques and kinematic analysis.

This study includes a prospective longitudinal study of patients with CP over one-year. This study will be executed in 3 phases within 3 years: 1st phase (1st years): to establish the multimodal brain images and motor control, and clinical outcomes protocol with a prospective one-year follow-up study in healthy subjects; 2nd phase (2nd years): to establish the brain images and motor control, and clinical outcomes with a prospective one-year follow-up study in older patients with CP; and 3rd phase (3rd years): to establish the brain images and motor control, and clinical outcomes with a prospective one-year follow-up study in younger patients with CP. In a prospective longitudinal study, each participant received 3-times measurements: at the beginning, 6 months later, and one year after the first data collection point

ELIGIBILITY:
Inclusion Criteria:

* (1) Age: 4-20 y/o (2) Good cognition and cooperation (3) Healthy participants

Exclusion Criteria:

* (1) Motor problems (2) Neurological, orthopedic, or progressive disorders (3) Active medical diseases, such as infection

Ages: 4 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: CP and healthy children
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2012-08; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline of functional magnetic resonance imaging (fMRI) analysis in 6 months and 12 months | baseline, 6 months, 12 months
  fc(functional connectivity)MRI at resting, active-task fMRI. diffusion tensor imaging (DTI)

SECONDARY OUTCOMES:
Change from baseline of kinematic analysis in 6 months and 12 months | baseline, 6 months, 12 months
  Kinematic analysis for upper limb and gait analysis
Change from baseline of movement and participation for Healthy children and CP in 6 months and 12 months | 6 months and 12 months
  Healthy children and CP: Bruininks- Oseretsky Test of Motor Proficiency II (BOT-2), Wolf Motor Function Test (WMFT), Block and Box test (BBT), Time up and go, Berg Balance Scale (BBS), Functional Independence Measure for Children (WeeFIM), Children Assessment of Participation and Enjoyment (CAPE), and School Function Assessment (SFA).
Change from baseline of movement and participation for CP in 6 months and 12 months | baseline, 6 months, 12 months
  Measures for CP also include Gross motor function measure (GMFM), Quality of upper extremity test (QUEST), Pediatric Motor Activity Log (PMAL), Caregiver Functional Use Survey (CFUS), etc.
Change from baseline of severity for CP patients in 6 months and 12 months | baseline, 6 months, 12 months
  CP patients: Gross Motor Functional Classification System (GMFCS), Manual Ability Classification System (MACS), Modified Ashworth Scale (MAS), strength and endurance, selective control, etc

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Ling Chen, PhD, Principal Investigator — Department of Physical Medicine & Rehabilitation, Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No